CLINICAL TRIAL: NCT03774511
Title: Effects of High-Intensity Interval and Moderate Intensity Continuous Exercise on Diabetic Obese Patients With Nonalcoholic Fatty Liver Disease- A Comparative Randomized Controlled Trial
Brief Title: Effects of Exercise on Patients With Nonalcoholic Fatty Liver Disease- A Comparative Randomized Controlled Trial
Acronym: [PTREC]
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ahlia University (Other)
Collaborators: Cairo University (Other)
Responsible Party: Principal Investigator, Dr Sayed Tantawy, Professor, Ahlia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T. REC/012/002146
Record Dates: First submitted 2018-12-12; First posted 2018-12-13 (Actual); Last update posted 2020-06-26 (Actual); Status verified 2020-06

CONDITIONS: Diabetes; Nonalcoholic Fatty Liver Disease; Obesity; Exercise
MeSH Terms: conditions — Diabetes Mellitus; Non-alcoholic Fatty Liver Disease; Obesity; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: HII group, each patient in this group were conducted a program of high-intensity aerobic exercise for 8 weeks, three times per week with each exercise session lasting for nearly 40 minutes morning. Each patient was instructed to not eat for 2 hours before the exercise session to avoid exercise induced airway obstruction. MIC group, each patient was received (MIC 3 times/week) for eight weeks, according to following parameters; 5 minutes warm up, followed by 30 minutes of continuous aerobic exercise on a cycle Ergometer with constant intensity at 70 to 75% of peak HR and 5 minutes cool down. Also, these measures were obtained at the beginning and the end of the intervention.
  Control group only received medical treatment with no exercise intervention
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Study group 1 (Active Comparator): High Intensity Interval Excercise
  Interventions: Other: High-Intensity Interval Exercise & Moderate Intensity Interval Exercise
- Study group 2 (Active Comparator): Moderate Intensity Interval Exercise
  Interventions: Other: High-Intensity Interval Exercise & Moderate Intensity Interval Exercise
- Control group (No Intervention): No Intervention

INTERVENTIONS:
Other: High-Intensity Interval Exercise & Moderate Intensity Interval Exercise — Different Interval intensities Exercise
  Other Names: Exercise
  Arms: Study group 1; Study group 2

SUMMARY:
background: Obesity, diabetes mellitus type II and fatty liver disease combining with low levels of physical activity are prominent health risks for mortality and morbidity. More than 1/3 of the current population is suffering from obesity with a significant proportion to medical complications which can negatively influence their quality of life. These complications comprise alterations of the metabolism of glucose and fat, insulin resistance and diabetes mellitus. Objectives The purpose of this study was to compare between high intensity interval exercise and moderate intensity continuous on diabetic obese patients with NAFLD. Methods: forty-seven diabetic obese individuals with NAFLD were enrolled in this study. The individuals were randomly divided into 16 in HII group, 15 in MIC group, and 16 in the controls. HII group received HII exercise, MIC group received 8-week MIC exercise while the control group did not receive any exercise intervention. IHTG and visceral lipids were assessed pre- and post-intervention.

DETAILED DESCRIPTION:
This randomized controlled trial initially included 48 diabetic obese patients with NAFLD, their age was 40 to 60 years and divide them equally into three groups. The data went to the analysis were 47 due to drop out of one subject. The 47 patients were randomly classified into 3 groups. Group I included 16 patients, received medical treatment with a program of HII exercise 3 times/wk for 8 weeks (HII group), group II included 15 patients, received moderate-intensity continuous (MIC) exercise 3 times/wk for 8 weeks (MIC group), and group III included 16 patients, received only medical treatment without exercise program (control).

Inclusion criteria: All patients were diagnosed with NAFLD, type II DM, and obesity (body mass index [BMI] ≥30 kg/m2). The diagnostic criteria of NAFLD based on the diagnostic guidelines for NAFLD in the Asia-Pacific region.[29] All study participants were non-smokers.

Exclusion criteria: Any patient had a severe life limiting illness (cancer, renal failure), uncontrolled heart disease, neuromuscular limitations, orthopedic problems, and endocrine disorders that could affect physical exercise was excluded from the study.

The HII exercise program was performed on a cycle Ergometer with firmly grasping the rails to maintain balance. The exercise session was started with a 5 minute warm up involving cycling exercise without resistance of the Ergometer followed by three sets of 4-min cycling sessions at 80-85% of the VO2max with 2-min interval at 50% of the VO2max between sets. The session was finished with 5 minutes of cool down exercise.

MIC group, each patient was received (MIC 3 times/week) for eight weeks, according to following parameters; 5 minutes warm up, followed by 30 minutes of continuous aerobic exercise on a cycle Ergometer with constant intensity at 70 to 75% of peak HR and 5 minutes cool down. Also, these measures were obtained at the beginning and the end of the intervention.

ELIGIBILITY:
Inclusion criteria:

* Clinical diagnosis of NAFLD, type II DM, and obesity.
* Body mass index (BMI) ≥30 kg/m2.
* Age: 40-60 years
* No smoking.

Exclusion criteria:

* Severe life limiting illness (cancer, renal failure),
* Uncontrolled heart disease,
* Neuromuscular limitations,
* Orthopedic problems
* Endocrine disorders that could affect physical exercise

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2017-07-09 (Actual); Primary Completion 2018-08-10 (Actual); Study Completion 2018-12-10 (Actual)

PRIMARY OUTCOMES:
Intrahepatic triglyceride (%) | 8 weeks
  Assessment in percentage (%) using MRI with a 3T scanner (General electric, WI) through imaging of chemical shift. Each patient was assessed for imaging in the supine position using the body coil. The patient was instructed to make a single breath hold during imaging, the liver was imaged 3 separate images slice pairs. IHTG proportionate to water was estimated as 100 × (signal amplitude of TG)/(signal amplitude of water).
Total cholesterol | 8 weeks
  Total cholesterol, (mg/dL)
Triglycerides | 8 weeks
  Triglycerides, (mg/dL)
High-density lipoproteins (HDLs) | 8 weeks
  High-density lipoproteins (HDLs), (mg/dL)
Low-density lipoproteins (LDLs) | 8 weeks
  Low-density lipoproteins (LDLs), (mg/dL)
Alanine-transaminase (ALT) | 8 weeks
  Alanine-transaminase (ALT), (IU/L)
Hemoglobin A1c (HbA1c) | 8 weeks
  Hemoglobin A1c (HbA1c), (%)
Homeostatic Model Assessment of Insulin Resistance (HOMA-IR) | 8 weeks
  It was assessed through Blood Code Calculation:
  HOMA-IR = Insulin (mU/L) х Glucose (mg/dL).

SECONDARY OUTCOMES:
Weight | 8 weeks
  Weight (kilograms Kg)
  * Alanine-transaminase (ALT), (IU/L)
  * Visceral adipose fat, (cm2) was assessed by MRI and anthropometric values.
  * Body mass index (BMI) in Kg/m2 was calculated as the weight (in kilograms) divided by height (in meters) squared.
Height | 8 weeks
  Height (meters m)
Body mass index (BMI) | 8 weeks
  Weight and height were combined to report BMI in kg/m^2
Visceral adipose fat | 8 weeks
  Visceral adipose fat, (cm2) was assessed by MRI and anthropometric values.

CONTACTS AND LOCATIONS:
Overall Officials: Sayed A Tantawy, PhD, Principal Investigator — Cairo University, Giza, Egypt; Walid K Abdelbasset, PhD, Study Director — Cairo University, Giza, Egypt
Locations (1):
- Dr Sayed Tanatwy, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No